CLINICAL TRIAL: NCT02424981
Title: Efficiency of Inspiratory Muscle Training in Elderly People
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Threshold IMT1
Record Dates: First submitted 2015-04-07; First posted 2015-04-23 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- inspiratory muscle training (Experimental): Muscle training
  Interventions: Device: Threshold inspiratory muscle training
- control (No Intervention): Control group

INTERVENTIONS:
Device: Threshold inspiratory muscle training — Inspiratory muscle training
  Arms: inspiratory muscle training

SUMMARY:
Efficiency of inspiratory muscle training in elderly people. Outcomes are lung function, muscle strength and chest expansion.

ELIGIBILITY:
Inclusion Criteria:

* healthy

Exclusion Criteria:

* pulmonary diseases
* cognitive disorders

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
lung function will be measured by spirometry | One month
chest expansion will be measured by a tape measure | One month

CONTACTS AND LOCATIONS:
Locations (1):
- Brussels, Belgium